CLINICAL TRIAL: NCT01106352
Title: A Phase I/IIa Study of Safety and Efficacy of Alpharadin® With Docetaxel in Patients With Bone Metastasis From Castration-Resistant Prostate Cancer
Brief Title: A Study of Alpharadin With Docetaxel in Patients With Bone Metastasis From Castration-Resistant Prostate Cancer (CRPC)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15469; BC1-10 (Other: Algeta ASA); 2011-000822-31 (EudraCT Number)
Record Dates: First submitted 2010-04-16; First posted 2010-04-19 (Estimated); Results first posted 2016-11-09 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2016-11

CONDITIONS: Bone Metastases; Castration-Resistant Prostate Cancer
Keywords: The target population is patients with bone metastasis from castration-resistant prostate cancer intended for treatment with docetaxel
MeSH Terms: interventions — radium Ra 223 dichloride; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Radium-223 dichloride (Xofigo, BAY88-8223) + docetaxel (Experimental): Alpharadin (Radium-223 dichloride) is administered intravenously as a bolus injection. In the randomized phase IIa part of the protocol, the dose established in the dose-escalation part of the protocol (Phase I) will be used, i.e. 5 doses of 50 kBq/kg b.w. every 6 weeks in combination with the approved step-down dose of docetaxel (60 mg/m^2) administered intravenously every 3 weeks with 5 mg prednisone twice a day continuously and pre-medication with dexamethasone.
  Interventions: Drug: Radium-223 dichloride (Xofigo, BAY88-8223); Drug: Docetaxel
- Docetaxel (Active Comparator): Docetaxel (75 mg/m2) will be administered intravenously every 3 weeks with 5 mg prednisone twice a day continuously and pre-medication with dexamethasone. Step-down to 60 mg/m^2 is allowed as per the approved docetaxel label.
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Radium-223 dichloride (Xofigo, BAY88-8223) — Alpharadin (Radium-223 dichloride) is administered intravenously as a bolus injection.
  Arms: Radium-223 dichloride (Xofigo, BAY88-8223) + docetaxel
Drug: Docetaxel — Docetaxel (75 mg/m^2) will be administered intravenously every 3 weeks with 5 mg prednisone twice a day continuously and pre-medication with dexamethasone. Step-down to 60 mg/m^2 is allowed as per the approved docetaxel label.

SUMMARY:
The main purpose of this study is to establish a recommended dose of Alpharadin to be used in combination with docetaxel in patients with bone metastases from castration-resistant prostate cancer and to investigate safety and explore efficacy of the recommended dose.

DETAILED DESCRIPTION:
The trial was initially conducted and submitted by Algeta ASA. After acquiring Algeta, Bayer is now the sponsor.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate.
* Two or more bone metastases (hot spots) confirmed by bone scintigraphy within 8 weeks prior to study entry
* Known castration-resistant disease
* Karnofsky Performance Status (KPS): ≥70% within 14 days before start of study treatment (ECOG 1)
* Life expectancy at least 6 months.
* Acceptable hematology and serum biochemistry screening values
* Eligible for use of docetaxel according to the product information (package insert or similar).

Exclusion Criteria:

* Has received an investigational therapeutic drug within the last 4 weeks prior to start of study treatment, or is scheduled to receive one during the treatment period.
* Has received external radiotherapy within the last 4 weeks prior to start of study treatment.
* Has an immediate need for radiotherapy.
* Has received prior hemibody external radiotherapy .
* Has received systemic radiotherapy (e.g. samarium, strontium etc.) for the treatment of bone metastases.
* Has received cytotoxic chemotherapy within the last 4 weeks prior to start of study treatment, or has not recovered to grade 1 or 0 from adverse events due to cytotoxic chemotherapy administered more than 4 weeks earlier.
* Has received more than ten previous infusions of docetaxel.
* Previous known experience of grade ≥ 3 docetaxel related toxicities or docetaxel toxicity related dose interruption or discontinuation.
* Previous use of G-CSF for persistent neutropenia after docetaxel treatment.
* Has received blood transfusion or erythropoietin (EPO) within the last 4 weeks prior to start of study treatment.
* Has received prior treatment with Alpharadin.
* Malignant lymphadenopathy exceeding 3 cm in short-axis diameter.
* Symptomatic nodal disease, i.e. scrotal, penile or leg edema.
* Visceral metastases from CRPC (>2 lung and/or liver metastases [size ≥2cm]), as assessed by CT scan or MRI of the chest/abdomen/pelvis within the last 8 weeks prior to start of study treatment.
* Uncontrolled loco-regional disease.
* Other primary tumor (other than CRPC) including haematological malignancy present within the last 5 years (except non-melanoma skin cancer or low-grade superficial bladder cancer).
* Has imminent or established spinal cord compression based on clinical findings and/or MRI.
* Unmanageable fecal incontinence

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2010-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (7):
- United States (6):
  - San Francisco, California
  - Evanston, Illinois
  - Baltimore, Maryland
  - Boston, Massachusetts
  - New York, New York
  - Seattle, Washington
- Villejuif, France

REFERENCES:
- [Derived] Morris MJ, Loriot Y, Sweeney CJ, Fizazi K, Ryan CJ, Shevrin DH, Antonarakis ES, Pandit-Taskar N, Deandreis D, Jacene HA, Vesselle H, Petrenciuc O, Lu C, Carrasquillo JA, Higano CS. Radium-223 in combination with docetaxel in patients with castration-resistant prostate cancer and bone metastases: a phase 1 dose escalation/randomised phase 2a trial. Eur J Cancer. 2019 Jun;114:107-116. doi: 10.1016/j.ejca.2019.04.007. Epub 2019 May 11. PMID 31082669
- [Derived] Gkialas IK, Fragkoulis C. Emerging therapies targeting castration-resistant prostate cancer. J BUON. 2015 Nov-Dec;20(6):1389-96. PMID 26854432
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at seven study centers in United States and one study center in France, between 23 July 2010 (first subject first visit) and 16 June 2015 (last subject last visit).
Pre-assignment Details: A total of 70 subjects were enrolled in the study. Of these 17 were in the dose escalation cohort in three dose groups of radium-223 and docetaxel. The remaining 53 subjects were in expanded safety cohort, of them 46 were dosed; 33 received a combination of radium-223 dichloride plus docetaxel and 13 subjects received docetaxel alone.
Groups:
- Alpharadin 25 kBq/kg + Docetaxel 75 mg/m^2 - Dose Escalation: Subjects received two intravenous injections of Alpharadin (Radium [Ra]-223 dichloride, BAY88-8223) at a dose of 25 kBq/kg body weight based on NIST 2010 standardization, separated by an interval of six weeks in combination with docetaxel at 75 mg/m^2 every three weeks; unless dose limiting toxicity (DLT) or other safety concerns limited the dose escalation.
- Alpharadin 25 kBq/kg + Docetaxel 60 mg/m^2 - Dose Escalation: Subjects received two intravenous injections of Alpharadin at a dose of 25 kBq/kg body weight based on NIST 2010 standardization, separated by an interval of six weeks in combination with docetaxel at 60 mg/m^2 every three weeks; unless DLT or other safety concerns limited the dose escalation.
- Alpharadin 50 kBq/kg + Docetaxel 60 mg/m^2 - Dose Escalation: Subjects received two intravenous injections of Alpharadin at a dose of 50 kBq/kg body weight based on NIST 2010 standardization, separated by an interval of six weeks in combination with docetaxel at 60 mg/m^2 every three weeks; unless DLT or other safety concerns limited the dose escalation.
- Alpharadin 50 kBq/kg + Docetaxel 60 mg/m^2 - Safety Cohort: Subjects received five intravenous injections of Alpharadin at a dose of 50 kBq/kg body weight based on NIST 2010 standardization, separated by an interval of six weeks in combination with docetaxel at 60 mg/m^2 every three weeks.
- Docetaxel 75 mg/m^2 - Safety Cohort: Subjects received docetaxel at 75 mg/m^2 twice daily every three weeks.
Period: Overall Study
Arm/Group | Alpharadin 25 kBq/kg + Docetaxel 75 mg/m^2 - Dose Escalation | Alpharadin 25 kBq/kg + Docetaxel 60 mg/m^2 - Dose Escalation | Alpharadin 50 kBq/kg + Docetaxel 60 mg/m^2 - Dose Escalation | Alpharadin 50 kBq/kg + Docetaxel 60 mg/m^2 - Safety Cohort | Docetaxel 75 mg/m^2 - Safety Cohort
Started | 7 | 3 | 7 | 36 | 17
Started Dose Escalation | 7 (Number of subjects for safety analysis set.) | 3 (Number of subjects for safety analysis set.) | 7 (Number of subjects for safety analysis set.) | 0 | 0
Completed Dose Escalation | 6 | 3 | 5 | 0 | 0
Started Safety Cohort | 0 | 0 | 0 | 36 | 17
Treated Safety Cohort | 0 | 0 | 0 | 33 (Number of subjects for safety analysis set.) | 13 (Number of subjects for safety analysis set.)
Completed Safety Cohort | 0 | 0 | 0 | 23 | 9
Completed | 6 | 3 | 5 | 23 (This group is only applicable for Safety cohort period.) | 9 (This group is only applicable for Safety cohort period.)
Not Completed | 1 | 0 | 2 | 13 | 8
Not completed — Subjects untreated | 0 | 0 | 0 | 3 | 4
Not completed — Sponsor Decision | 1 | 0 | 0 | 0 | 0
Not completed — Too ill to come in for the visit | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 1 | 3 | 1
Not completed — Disease progression | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 3 | 2
Not completed — Went on hospice | 0 | 0 | 0 | 1 | 0
Not completed — Subject entered hospice | 0 | 0 | 0 | 1 | 0
Not completed — Home hospice since July 2013 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alpharadin 25 kBq/kg + Docetaxel 75 mg/m^2 - Dose Escalation | Alpharadin 25 kBq/kg + Docetaxel 60 mg/m^2 - Dose Escalation | Alpharadin 50 kBq/kg + Docetaxel 60 mg/m^2 - Dose Escalation | Alpharadin 50 kBq/kg + Docetaxel 60 mg/m^2 - Safety Cohort | Docetaxel 75 mg/m^2 - Safety Cohort | Total
Number analyzed (Participants) | 7 | 3 | 7 | 36 | 17 | 70
Age, Customized [Number; unit: participants]
  <18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 3 | 11 | 7 | 25
  >65 years | 5 | 1 | 4 | 25 | 10 | 45
Gender [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 7 | 3 | 7 | 36 | 17 | 70

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Dose-Limiting Toxicities - Dose Escalation Part
Description: DLT was defined as - Absolute neutrophil count grade greater than or equal to (>=) 4 (Common Terminology Criteria for Adverse Events [CTCAE], Version 4.0: less than [<] 0.5 × 109 per Liter) lasting longer than 7 days without fever despite granulocyte colony-stimulating factor (G-CSF) support). Platelet count Grade >= 4 (CTCAE, v4.0: < 25× 109/L) lasting longer than 7 days. Diarrhea Grade >= 3 (CTAE, v4.0: increase of >= 7 stools per day over baseline; incontinence; hospitalization indicated; severe increase in ostomy output compared with baseline; limiting self-care in activities of daily living) in spite of optimal use of antidiarrheal medication. Vomiting or constipation Grade >= 4 (CTCAE, v4.0: life-threatening consequences; urgent intervention indicated). Febrile neutropenia Grade >= 3 (CTCAE, v4.0).
Time Frame: From randomization until 6 weeks post-injection in all dose cohort of dose-escalation part
Measure: Number; unit: Participants
Arm/Group | Alpharadin 25 kBq/kg + Docetaxel 75 mg/m^2 - Dose Escalation | Alpharadin 25 kBq/kg + Docetaxel 60 mg/m^2 - Dose Escalation | Alpharadin 50 kBq/kg + Docetaxel 60 mg/m^2 - Dose Escalation
Number analyzed (Participants) | 7 | 3 | 7
Participants | 0 | 0 | 0

2. Primary Outcome: Number of Subjects With Treatment-Emergent Adverse Events (TEAE), Treatment-Emergent Serious Adverse Events (TESAE) With a CTCAE Grade of 3 or 4
Description: Treatment-emergent adverse event (TEAEs) were defined as events that occur following the first injection of study treatment, or that started prior to the first injection and worsened during treatment. An adverse event (AE) was any untoward medical occurrence in a subject who received study drug without regard to possibility of causal relationship. An Serious Adverse Event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged in patient hospitalization; lifethreatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent adverse events were defined as adverse events/serious adverse events that started or worsened after the study drug treatment.
Time Frame: From start of study treatment to 6 weeks after study treatment (that is maximum 12 weeks in dose escalation; 30 weeks in the expanded safety cohort) and 8 weeks for serious AEs
Population: Only participants who received treatment were assessed
Measure: Number; unit: Participants
Arm/Group | Alpharadin 25 kBq/kg + Docetaxel 75 mg/m^2 - Dose Escalation | Alpharadin 25 kBq/kg + Docetaxel 60 mg/m^2 - Dose Escalation | Alpharadin 50 kBq/kg + Docetaxel 60 mg/m^2 - Dose Escalation | Alpharadin 50 kBq/kg + Docetaxel 60 mg/m^2 - Safety Cohort | Docetaxel 75 mg/m^2 - Safety Cohort
Number analyzed (Participants) | 7 | 3 | 7 | 33 | 13
Participants
  TEAE CTCAE Grade 3 | 3 | 1 | 4 | 6 | 3
  TEAE CTCAE Grade 4 | 2 | 1 | 1 | 10 | 6
  TESAE | 4 | 0 | 2 | 7 | 4

3. Primary Outcome: Change From Baseline in Serum Biochemistry (Albumin, Protein, Hemoglobin) During the Treatment Period
Description: In the below table, 'n' signifies those subjects who were evaluable for this measure at given time points for each group.
Time Frame: Baseline, Day 106 (dose escalation period), and Day 190 (expanded safety cohort)
Population: Only randomized participants who have this outcome measure tested were assessed
Measure: Mean (Standard Deviation); unit: gram per liter (G/L)
Arm/Group | Alpharadin 25 kBq/kg + Docetaxel 75 mg/m^2 - Dose Escalation | Alpharadin 25 kBq/kg + Docetaxel 60 mg/m^2 - Dose Escalation | Alpharadin 50 kBq/kg + Docetaxel 60 mg/m^2 - Dose Escalation | Alpharadin 50 kBq/kg + Docetaxel 60 mg/m^2 - Safety Cohort | Docetaxel 75 mg/m^2 - Safety Cohort
Number analyzed (Participants) | 7 | 3 | 7 | 35 | 13
gram per liter (G/L)
  Albumin Baseline (n= 7,3,7,35,13) | 42 (3) | 43 (4) | 43 (3.56) | 42.7 (3.25) | 42.3 (4.09)
  Albumin: Change at Day 106 (n=1,0,0,27,11) | -2 (NA) — Standard deviation is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | -1.3 (2.98) | -1.2 (2.75)
  Albumin: Change at Day 190 (n= 0,0,0,24,6) | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | -2.3 (3.33) | -0.5 (2.07)
  Protein: Baseline (n= 7,3,7,35,13) | 70.3 (4.23) | 69.7 (8.5) | 70.4 (4.89) | 68.7 (4.45) | 69.1 (5.33)
  Protein: Change at Day 106 (n=1,0,0,27,11 ) | 1 (NA) — Standard deviation is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | -3.9 (3.79) | -3.8 (2.56)
  Protein: Change at Day 190 (n= 0,0,0,24,6) | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | -5.3 (3.63) | -3.7 (4.18)
  Hemoglobin: Baseline (n= 7,3,7,35,13) | 122.43 (14.581) | 120.67 (16.166) | 120.43 (8.522) | 122.82 (10.939) | 120.23 (12.05)
  Hemoglobin: Change at Day 106 (n=1,0,0,27,11 ) | -10 (NA) — Standard deviation is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | -8.81 (8.2) | -14.27 (9.067)
  Hemoglobin: Change at Day 190 (n= 0,0,0,23,6) | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | -13.65 (10.853) | -10.67 (13.794)

4. Primary Outcome: Change From Baseline in Serum Biochemistry (Alkaline Phosphatase [AP], Alanine Aminotransferase [AAT], Lactate Dehydrogenase [LD]) During the Treatment Period
Description: as for outcome 3
Time Frame: Baseline, Day 106 (dose escalation period), and Day 190 (expanded safety cohort)
Population: Only participants who received treatment were assessed
Measure: Mean (Standard Deviation); unit: units per liter (U/L)
Arm/Group | Alpharadin 25 kBq/kg + Docetaxel 75 mg/m^2 - Dose Escalation | Alpharadin 25 kBq/kg + Docetaxel 60 mg/m^2 - Dose Escalation | Alpharadin 50 kBq/kg + Docetaxel 60 mg/m^2 - Dose Escalation | Alpharadin 50 kBq/kg + Docetaxel 60 mg/m^2 - Safety Cohort | Docetaxel 75 mg/m^2 - Safety Cohort
Number analyzed (Participants) | 7 | 3 | 7 | 33 | 17
units per liter (U/L)
  AP: Baseline (n= 7,3,7,33,13) | 533.1 (656.36) | 144 (89.2) | 224.6 (115.08) | 218.2 (207.63) | 195.9 (110.86)
  AP: Change at Day 106 (n=1,0,0,27,11) | -134 (NA) — Standard deviation is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | -119.6 (153.1) | -78.9 (46.35)
  AP: Change at Day 190 (n= 0,0,0,24,6) | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | -119.3 (112.21) | -116.8 (52.21)
  AAT: Baseline (n= 7,3,7,33,13) | 17.6 (5.68) | 17 (6.56) | 18.9 (5.9) | 19.8 (9.82) | 19.8 (10.78)
  AAT: Change at Day 106 (n=1,0,0,27,11 ) | 100 (NA) — Standard deviation is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | 2.9 (13.54) | -2.2 (11.75)
  AAT: Change at Day 190 (n= 0,0,0,24,6) | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | 1.1 (8.67) | -3.7 (13.81)
  LD: Baseline (n= 7,3,7,33,13) | 313.3 (243.9) | 179 (22.52) | 214.4 (38.92) | 212.8 (71.07) | 203.4 (61.68)
  LD: Change at Day 106 (n= 1,0,0,27,11) | 15 (NA) — Standard deviation is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | 10.7 (58.14) | 45.1 (93.58)
  LD: Change at Day 190 (n= 0,0,0,24,6) | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | 16.9 (39.74) | 17.5 (100.85)

5. Primary Outcome: Change From Baseline in Serum Biochemistry (Bilirubin, Creatinine) During the Treatment Period
Description: as for outcome 3
Time Frame: Baseline, Day 106 (dose escalation period), and Day 190 (expanded safety cohort)
Population: Only participants who received treatment were assessed
Measure: Mean (Standard Deviation); unit: micromole(s)/litre
Arm/Group | Alpharadin 25 kBq/kg + Docetaxel 75 mg/m^2 - Dose Escalation | Alpharadin 25 kBq/kg + Docetaxel 60 mg/m^2 - Dose Escalation | Alpharadin 50 kBq/kg + Docetaxel 60 mg/m^2 - Dose Escalation | Alpharadin 50 kBq/kg + Docetaxel 60 mg/m^2 - Safety Cohort | Docetaxel 75 mg/m^2 - Safety Cohort
Number analyzed (Participants) | 7 | 3 | 7 | 33 | 13
micromole(s)/litre
  Bilirubin: Baseline (n= 7,3,7,33,13) | 8.9 (3.8) | 6.7 (1.15) | 7.1 (3.98) | 7.5 (2.62) | 7 (2.08)
  Bilirubin: Change at Day 106 (n= 1,0,0,27,11) | 2 (NA) — Standard deviation is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | 0.2 (1.84) | -0.8 (1.72)
  Bilirubin: Change at Day 190 (n= 0,0,0,24,6) | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | -0.9 (1.56) | 0.3 (1.51)
  Creatinine: Baseline (n= 7,3,7,33,13) | 92.33 (33.126) | 73.67 (9.5) | 70.86 (10.938) | 70.07 (19.138) | 75.5 (11.614)
  Creatinine: Change at Day 106 (n= 1,0,0,27,11) | 63.6 (NA) — Standard deviation is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | 0.74 (12.273) | -0.7 (7.232)
  Creatinine: Change at Day 190 (n= 0,0,0,24,6) | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | 0.59 (11.889) | -0.17 (13.31)

6. Primary Outcome: Change From Baseline in Serum Biochemistry (Calcium, Chloride, Magnesium, Potassium, Phosphate, Sodium, Urea) During the Treatment Period
Description: as for outcome 3
Time Frame: Baseline, Day 106 (dose escalation period), and Day 190 (expanded safety cohort)
Population: Only participants who received treatment were assessed
Measure: Mean (Standard Deviation); unit: millimole(s)/liter
Arm/Group | Alpharadin 25 kBq/kg + Docetaxel 75 mg/m^2 - Dose Escalation | Alpharadin 25 kBq/kg + Docetaxel 60 mg/m^2 - Dose Escalation | Alpharadin 50 kBq/kg + Docetaxel 60 mg/m^2 - Dose Escalation | Alpharadin 50 kBq/kg + Docetaxel 60 mg/m^2 - Safety Cohort | Docetaxel 75 mg/m^2 - Safety Cohort
Number analyzed (Participants) | 7 | 3 | 7 | 33 | 13
millimole(s)/liter
  Calcium: Baseline (n= 7,3,7,33,13) | 2.231 (0.1523) | 2.38 (0.0872) | 2.309 (0.071) | 2.357 (0.1121) | 2.307 (0.1437)
  Calcium: Change at Day 106 (n= 1,0,0,27,11) | 0.2 (NA) — Standard deviation is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | -0.065 (0.148) | -0.019 (0.104)
  Calcium: Change at Day 190 (n= 0,0,0,24,6) | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | -0.055 (0.1225) | -0.143 (0.1536)
  Chloride: Baseline (n= 7,3,7,33,13) | 101.4 (3.21) | 101.7 (2.52) | 102 (2.77) | 103.2 (2.75) | 101.3 (3.99)
  Chloride: Change at Day 106 (n= 1,0,0,27,11) | -1.9 (NA) — Standard deviation is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | 0 (2.72) | 1.5 (2.38)
  Chloride: Change at Day 190 (n= 0,0,0,24,6) | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | 0 (3.35) | 2.5 (1.38)
  Magnesium: Baseline (n= 7,3,7,33,13) | 0.93 (0.055) | 0.86 (0) | 0.86 (0.088) | 0.85 (0.072) | 0.84 (0.073)
  Magnesium: Change at Day 106 (n= 1,0,0,27,11) | -4.4 (NA) — Standard deviation is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | -0.02 (0.058) | -0.04 (0.036)
  Magnesium: Change at Day 190 (n= 0,0,0,24,6) | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | -0.01 (0.079) | -0.06 (0.045)
  Potassium: Baseline (n= 7,3,7,33,13) | 4.34 (0.541) | 4.47 (0.306) | 4.39 (0.09) | 4.29 (0.277) | 4.3 (0.443)
  Potassium: Change at Day 106 (n= 1,0,0,27,11) | 1.1 (NA) — Standard deviation is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | 0.06 (0.366) | 0.11 (0.336)
  Potassium: Change at Day 190 (n= 0,0,0,24,6) | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | 0.04 (0.422) | 0.03 (0.501)
  Phosphate: Baseline (n= 7,3,7,33,13) | 1.021 (0.168) | 1.167 (0.2466) | 0.993 (0.369) | 1.058 (0.1763) | 1.145 (0.1844)
  Phosphate: Change at Day 106 (n= 1,0,0,27,11) | 0 (NA) — Standard deviation is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | 0.086 (0.1369) | -0.061 (0.2287)
  Phosphate: Change at Day 190 (n= 0,0,0,24,6) | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | 0.128 (0.1734) | 0.203 (0.1813)
  Sodium: Baseline (n= 7,3,7,33,13) | 136.1 (4.1) | 137.7 (3.51) | 137.4 (2.51) | 138.5 (2.49) | 137.2 (4.72)
  Sodium: Change at Day 106 (n= 1,0,0,27,11) | 0 (NA) — Standard deviation is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | -0.6 (2.28) | 0.8 (2.56)
  Sodium: Change at Day 190 (n= 0,0,0,24,6) | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | -0.5 (2.41) | 2.3 (1.37)
  Urea: Baseline (n= 7,3,7,33,13) | 9.14 (3.092) | 7.83 (1.041) | 6.79 (2.059) | 7.03 (2.304) | 7.78 (2.312)
  Urea: Change at Day 106 (n= 1,0,0,27,11) | 1.5 (NA) — Standard deviation is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | -0.26 (1.587) | -0.26 (1.531)
  Urea: Change at Day 190 (n= 0,0,0,24,6) | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | -0.15 (1.508) | 0.7 (1.122)

7. Primary Outcome: Change From Baseline in Serum Biochemistry (Platelets, Leukocytes, Lymphocytes, Neutrophils, Monocytes, Eosinophils, Basophils) During the Treatment Period
Description: as for outcome 3
Time Frame: Baseline, Day 106 (dose escalation period), and Day 190 (expanded safety cohort)
Population: Only participants who received treatment were assessed
Measure: Mean (Standard Deviation); unit: giga per liter (GI/L)
Arm/Group | Alpharadin 25 kBq/kg + Docetaxel 75 mg/m^2 - Dose Escalation | Alpharadin 25 kBq/kg + Docetaxel 60 mg/m^2 - Dose Escalation | Alpharadin 50 kBq/kg + Docetaxel 60 mg/m^2 - Dose Escalation | Alpharadin 50 kBq/kg + Docetaxel 60 mg/m^2 - Safety Cohort | Docetaxel 75 mg/m^2 - Safety Cohort
Number analyzed (Participants) | 7 | 3 | 7 | 33 | 13
giga per liter (GI/L)
  Platelets: Baseline (n= 7,3,7,33,13) | 214.1 (58.05) | 196.3 (51.64) | 266.6 (77.43) | 259.6 (69.39) | 240.6 (52.17)
  Platelets: Change at Day 106 (n= 1,0,0,27,11) | 169 (NA) — Standard deviation is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | -3.1 (51.39) | 33 (55.17)
  Platelets: Change at Day 190 (n= 0,0,0,23,6) | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | -22 (51.04) | 32.3 (68.54)
  Leukocytes: Baseline (n= 7,3,7,33,13) | 9.13 (4.43) | 5.83 (1.858) | 8.34 (2.783) | 7.67 (2.871) | 6.71 (2.308)
  Leukocytes: Change at Day 106 (n= 1,0,0,27,11) | 18.7 (NA) — Standard deviation is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | -0.1 (2.086) | 2.44 (2.263)
  Leukocytes: Change at Day 190 (n= 0,0,0,23,6) | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | -0.12 (2.603) | 1.65 (1.946)
  Lymphocytes: Baseline (n= 7,3,7,33,13) | 1.044 (0.4687) | 1.003 (0.45) | 0.81 (0.4679) | 1.001 (0.5902) | 1.068 (0.5751)
  Lymphocytes: Change at Day 106 (n= 1,0,0,27,11) | 1.3 (NA) — Standard deviation is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | -0.229 (0.5593) | -0.063 (0.5129)
  Lymphocytes: Change at Day 190 (n= 0,0,0,23,6) | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | -0.395 (0.3917) | -0.085 (0.6832)
  Neutrophils: Baseline (n= 7,3,7,33,13) | 7.809 (4.0998) | 4.71 (1.54) | 7.359 (2.7781) | 6.363 (2.8618) | 5.205 (2.1487)
  Neutrophils: Change at Day 106 (n= 1,0,0,27,11) | 517.3 (NA) — Standard deviation is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | 0.178 (2.2991) | 2.622 (2.5672)
  Neutrophils: Change at Day 190 (n= 0,0,0,23,6) | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | 0.341 (2.4734) | 2.038 (1.8799)
  Monocytes: Baseline (n= 7,3,7,33,13) | 0.224 (0.2319) | 0.103 (0.085) | 0.153 (0.1379) | 0.243 (0.2466) | 0.375 (0.4203)
  Monocytes: Change at Day 106 (n= 1,0,0,27,11) | 0.12 (NA) — Standard deviation is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | -0.011 (0.2959) | -0.111 (0.4164)
  Monocytes: Change at Day 190 (n= 0,0,0,23,6) | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | -0.014 (0.3185) | -0.27 (0.2964)
  Eosinophils: Baseline (n= 7,3,7,33,13) | 0.04 (0.0622) | 0.01 (0.01) | 0.014 (0.0151) | 0.054 (0.0734) | 0.043 (0.0407)
  Eosinophils: Change at Day 106 (n= 1,0,0,27,11) | -0.12 (NA) — Standard deviation is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | -0.043 (0.0797) | -0.008 (0.0995)
  Eosinophils: Change at Day 190 (n= 0,0,0,23,6) | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | -0.049 (0.0786) | -0.023 (0.0186)
  Basophils: Baseline (n= 7,3,7,33,13) | 0.013 (0.0221) | 0.007 (0.0058) | 0.011 (0.0107) | 0.012 (0.0137) | 0.018 (0.0121)
  Basophils: Change at Day 106 (n= 1,0,0,27,11) | 0.02 (NA) — Standard deviation is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | 0.001 (0.0169) | -0.001 (0.0197)
  Basophils: Change at Day 190 (n= 0,0,0,23,6) | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | -0.003 (0.0136) | -0.015 (0.0105)

8. Primary Outcome: Change From Baseline in Serum Biochemistry (Erythrocytes) During the Treatment Period
Description: as for outcome 3
Time Frame: Baseline, Day 106 (dose escalation period), and Day 190 (expanded safety cohort)
Population: Only participants who received treatment were assessed
Measure: Mean (Standard Deviation); unit: tetra per liter (TI/L)
Arm/Group | Alpharadin 25 kBq/kg + Docetaxel 75 mg/m^2 - Dose Escalation | Alpharadin 25 kBq/kg + Docetaxel 60 mg/m^2 - Dose Escalation | Alpharadin 50 kBq/kg + Docetaxel 60 mg/m^2 - Dose Escalation | Alpharadin 50 kBq/kg + Docetaxel 60 mg/m^2 - Safety Cohort | Docetaxel 75 mg/m^2 - Safety Cohort
Number analyzed (Participants) | 7 | 3 | 7 | 33 | 13
tetra per liter (TI/L)
  Erythrocytes: Baseline (n= 7,3,7,33,13) | 3.99 (0.376) | 3.9 (0.361) | 3.9 (0.327) | 3.98 (0.378) | 4.02 (0.519)
  Erythrocytes: Change at Day 106 (n= 1,0,0,27,11) | -0.4 (NA) — Standard deviation is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | -0.25 (0.233) | -0.32 (0.429)
  Erythrocytes: Change at Day 190 (n= 0,0,0,23,6) | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | -0.39 (0.287) | -0.15 (0.653)

9. Primary Outcome: Changes From Baseline in Systolic and Diastolic Blood Pressure During the Treatment Period
Description: as for outcome 3
Time Frame: From start of study treatment to 6 weeks after study treatment (that is, maximum 12 weeks in dose escalation; 30 weeks in the expanded safety cohort)
Population: Only participants who received treatment were assessed
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Alpharadin 25 kBq/kg + Docetaxel 75 mg/m^2 - Dose Escalation | Alpharadin 25 kBq/kg + Docetaxel 60 mg/m^2 - Dose Escalation | Alpharadin 50 kBq/kg + Docetaxel 60 mg/m^2 - Dose Escalation | Alpharadin 50 kBq/kg + Docetaxel 60 mg/m^2 - Safety Cohort | Docetaxel 75 mg/m^2 - Safety Cohort
Number analyzed (Participants) | 7 | 3 | 7 | 33 | 13
millimeters of mercury (mmHg)
  SBP: Baseline (n= 7,3,7,33,13) | 137.7 (9.11) | 113 (12.12) | 131.7 (13.07) | 139.2 (17.01) | 140.1 (10.85)
  SBP: Change at Day 22 (n= 6,3,7,33,13) | -2.7 (13.52) | 2.3 (5.51) | -5 (12.32) | -1.8 (19.66) | -8.5 (19.53)
  SBP: Change at Day 43 (n= 6,3,7,32,13) | -8.7 (12.13) | -3 (9.54) | -0.9 (19.37) | 0.6 (18.15) | -15.3 (13.91)
  SBP: Change at Day 64 (n= 6,3,6,30,13) | -9.8 (16.36) | -11 (13.45) | -4.2 (13.66) | -2.5 (21.75) | -10.1 (13.32)
  SBP: Change at Day 85 (n= 0,0,0,28,13) | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | -3.1 (16.55) | -3.8 (17.19)
  SBP: Change at Day 106 (n= 0,0,0,28,12) | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | -6.7 (21.33) | -10.4 (16.33)
  SBP: Change at Day 127 (n= 0,0,0,27,8) | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | -4.6 (19.82) | -13.4 (22.01)
  SBP: Change at Day 148 (n= 0,0,0,25,7) | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | -3.9 (20.09) | -8.9 (18.02)
  SBP: Change at Day 169 (n= 0,0,0,25,7) | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | -3.6 (16.58) | -6.3 (17.85)
  SBP: Change at Day 190 (n= 0,0,0,24,6) | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | -8.1 (18.25) | -10 (16.15)
  DBP: Baseline (n= 7,3,7,33,13) | 81.6 (5.68) | 62 (2) | 74.1 (8.86) | 76.1 (10.19) | 83 (11.17)
  DBP: Change at Day 22 (n= 6,3,7,33,13) | -2.7 (10.67) | 8 (10.39) | 2.6 (7.57) | 0.3 (10.88) | -6.2 (16.03)
  DBP: Change at Day 43 (n= 6,3,7,32,13) | -3.7 (6.65) | 2.7 (5.03) | 4.1 (8.13) | -1.8 (12.17) | -11.7 (10.89)
  DBP: Change at Day 64 (n= 6,3,6,30,13) | -8.7 (7.89) | -1 (1.73) | -0.2 (15.93) | -1.4 (14.66) | -8.7 (9.21)
  DBP: Change at Day 85 (n= 0,0,0,28,13) | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | 1.1 (10.99) | -7.6 (11.2)
  DBP: Change at Day 106 (n= 0,0,0,28,12) | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | -0.8 (13.15) | -7.9 (14.13)
  DBP: Change at Day 127 (n= 0,0,0,27,8) | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | -1.4 (14.22) | -8 (9.94)
  DBP: Change at Day 148 (n= 0,0,0,25,7) | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | -2 (12.19) | -3.9 (8.36)
  DBP: Change at Day 169 (n= 0,0,0,25,7) | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | -1.2 (10.45) | -9 (8.6)
  DBP: Change at Day 190 (n= 0,0,0,24,6) | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | -3.6 (12.8) | -12 (8.92)

10. Primary Outcome: Changes From Baseline in Respiratory Rate During the Treatment Period
Description: as for outcome 3
Time Frame: as for outcome 9
Population: Only participants who received treatment were assessed
Measure: Mean (Standard Deviation); unit: breaths/min
Arm/Group | Alpharadin 50 kBq/kg + Docetaxel 60 mg/m^2 - Dose Escalation | Alpharadin 25 kBq/kg + Docetaxel 60 mg/m^2 - Dose Escalation | Alpharadin 25 kBq/kg + Docetaxel 75 mg/m^2 - Dose Escalation | Alpharadin 50 kBq/kg + Docetaxel 60 mg/m^2 - Safety Cohort | Docetaxel 75 mg/m^2 - Safety Cohort
Number analyzed (Participants) | 7 | 3 | 7 | 33 | 13
breaths/min
  Baseline (n= 7,3,7,33,13) | 19.3 (1.63) | 18.7 (2.31) | 19.1 (1.57) | 17.1 (2.67) | 17.5 (2.79)
  Change at Day 22 (n= 6,3,7,33,13) | -1.7 (2.34) | -1.3 (2.31) | -0.7 (1.03) | 0.3 (2.1) | -0.4 (2.14)
  Change at Day 43 (n= 6,3,7,32,13) | 0 (1.26) | 1.3 (4.62) | -0.3 (0.82) | 0 (3.08) | 0.7 (3.5)
  Change at Day 64 (n= 6,3,6,30,13) | -0.5 (2.81) | 0 (4) | -1 (1.1) | 0.4 (2.82) | 0.8 (3)
  Change at Day 85 (n= 0,0,0,28,13) | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | 0 (3.32) | -0.3 (2.39)
  Change at Day 106 (n= 0,0,0,28,12) | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | -0.8 (3.54) | 0.5 (3.27)
  Change at Day 127 (n= 0,0,0,27,8) | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | 0.9 (3.69) | 0.4 (1.51)
  Change at Day 148 (n= 0,0,0,25,7) | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | 0.7 (3.38) | -0.3 (1.51)
  Change at Day 169 (n= 0,0,0,25,7) | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | -1 (3.11) | 0.4 (2.15)
  Change at Day 190 (n= 0,0,0,24,6) | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | 0 (4.79) | -0.2 (1.33)

11. Primary Outcome: Changes From Baseline in Heart Rate During the Treatment Period
Description: as for outcome 3
Time Frame: as for outcome 9
Population: Only participants who received treatment were assessed
Measure: Mean (Standard Deviation); unit: beats per min
Arm/Group | Alpharadin 25 kBq/kg + Docetaxel 75 mg/m^2 - Dose Escalation | Alpharadin 25 kBq/kg + Docetaxel 60 mg/m^2 - Dose Escalation | Alpharadin 50 kBq/kg + Docetaxel 60 mg/m^2 - Dose Escalation | Alpharadin 50 kBq/kg + Docetaxel 60 mg/m^2 - Safety Cohort | Docetaxel 75 mg/m^2 - Safety Cohort
Number analyzed (Participants) | 7 | 3 | 7 | 33 | 13
beats per min
  Baseline (n= 7,3,7,33,13) | 88.6 (18.84) | 58 (9.17) | 80 (9.93) | 77.9 (14.18) | 73.3 (12.01)
  Change at Day 22 (n= 6,3,7,33,13) | -0.2 (6.49) | 9.7 (18.72) | -0.6 (7.76) | 2 (11.39) | 7.2 (12.17)
  Change at Day 43 (n= 6,3,7,32,13) | -4.3 (9.35) | 18.3 (14.57) | 0.9 (10.32) | 2.8 (11.13) | 4.9 (11.54)
  Change at Day 64 (n= 6,3,6,30,13) | 0.7 (7.28) | 13 (21.17) | 6.5 (11.47) | 3.4 (14.48) | 5.1 (9.41)
  Change at Day 85 (n= 0,0,0,28,13) | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | 2.9 (16.17) | 7.2 (10.27)
  Change at Day 106 (n= 0,0,0,28,12) | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | 0.8 (19.18) | 9.2 (11.67)
  Change at Day 127 (n= 0,0,0,27,8) | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | 2.2 (13.93) | 7.5 (5.86)
  Change at Day 148 (n= 0,0,0,25,7) | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | 2.2 (15.88) | 15.3 (14.38)
  Change at Day 169 (n= 0,0,0,25,7) | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | 3.6 (16.91) | 8 (7.72)
  Change at Day 190 (n= 0,0,0,24,6) | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | 2.6 (16.01) | 18 (11.31)

12. Primary Outcome: Changes From Baseline in Weight During the Treatment Period
Description: as for outcome 3
Time Frame: as for outcome 9
Population: Only participants who received treatment were assessed
Measure: Mean (Standard Deviation); unit: kilogram(s)
Arm/Group | Alpharadin 25 kBq/kg + Docetaxel 75 mg/m^2 - Dose Escalation | Alpharadin 25 kBq/kg + Docetaxel 60 mg/m^2 - Dose Escalation | Alpharadin 50 kBq/kg + Docetaxel 60 mg/m^2 - Dose Escalation | Alpharadin 50 kBq/kg + Docetaxel 60 mg/m^2 - Safety Cohort | Docetaxel 75 mg/m^2 - Safety Cohort
Number analyzed (Participants) | 7 | 3 | 7 | 33 | 13
kilogram(s)
  Baseline (n= 7,3,7,33,13) | 89.3 (13.15) | 81.9 (21.66) | 97.1 (14.29) | 87.7 (14.81) | 92 (22.28)
  Change at Day 22 (n= 6,3,7,33,13) | -1.8 (1.31) | -0.3 (1.55) | -1.4 (2.5) | -0.4 (1.42) | -0.2 (1.92)
  Change at Day 43 (n= 6,3,7,32,13) | -1 (1.95) | 0.2 (2.2) | -1 (2.99) | 0 (2.2) | 0.5 (1.98)
  Change at Day 64 (n= 6,3,6,30,13) | 0.1 (4.2) | 0.3 (2.04) | -1.2 (3.08) | 0.2 (2.41) | 0.3 (2.48)
  Change at Day 85 (n= 0,0,0,28,13) | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | -0.2 (3.47) | 0.4 (2.87)
  Change at Day 106 (n= 0,0,0,28,12) | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | -0.3 (3.53) | 0.4 (3.1)
  Change at Day 127 (n= 0,0,0,27,8) | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | -0.1 (4.09) | 2.1 (2.11)
  Change at Day 148 (n= 0,0,0,25,7) | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | -0.1 (4.45) | 1.9 (2.72)
  Change at Day 169 (n= 0,0,0,25,7) | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | -0.1 (4.53) | 1.7 (3.81)
  Change at Day 190 (n= 0,0,0,24,6) | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | NA (NA) — Mean Value is not calculated. | 0.1 (5) | -0.7 (3.59)

13. Primary Outcome: Number of Subjects With Physical Examination During the Treatment Period
Description: Any physical examination finding that was classified by the investigator as a clinically significant change (compared with previous examination) was considered an AE, documented on the eCRF, and followed until the outcome was known. The below physical examination findings were recorded and reported. GDASC = General disorders and administration site conditions MND = Metabolism and nutrition disorders SSTD= Skin and subcutaneous tissue disorders MCTD = Musculoskeletal and connective tissue disorders IPPC = Injury, poisoning and procedural complications RTMD = Respiratory, thoracic and mediastinal disorders NBMU = Neoplasms benign, malignant and unspecified (include cysts and polyps) In the below table.
Time Frame: From start of study treatment to 6 weeks after study treatment (i.e., maximum 12 weeks in dose escalation; 30 weeks in the expanded safety cohort)
Population: Only participants who received treatment were assessed
Measure: Number; unit: Participants
Arm/Group | Alpharadin 25 kBq/kg + Docetaxel 75 mg/m^2 - Dose Escalation | Alpharadin 25 kBq/kg + Docetaxel 60 mg/m^2 - Dose Escalation | Alpharadin 50 kBq/kg + Docetaxel 60 mg/m^2 - Dose Escalation | Alpharadin 50 kBq/kg + Docetaxel 60 mg/m^2 - Safety Cohort | Docetaxel 75 mg/m^2 - Safety Cohort
Number analyzed (Participants) | 7 | 3 | 7 | 33 | 13
Participants
  At day 64: GDASC | 0 | 0 | 2 | 5 | 2
  At day 64: MND | NA — Data was not collected. | NA — Data was not collected. | NA — Data was not collected. | 0 | 1
  At day 64: SSTD | NA — Data was not collected. | NA — Data was not collected. | NA — Data was not collected. | 2 | 6
  At day 190: GDASC | NA — The time frame is only applicable to safety cohort. | NA — The time frame is only applicable to safety cohort. | NA — The time frame is only applicable to safety cohort. | 7 | 2
  At day 190: MCTD | NA — The time frame is only applicable to safety cohort. | NA — The time frame is only applicable to safety cohort. | NA — The time frame is only applicable to safety cohort. | 1 | 0
  At day 190: SSTD | NA — The time frame is only applicable to safety cohort. | NA — The time frame is only applicable to safety cohort. | NA — The time frame is only applicable to safety cohort. | 7 | 2
  At day 190: Vascular disorders | NA — The time frame is only applicable to safety cohort. | NA — The time frame is only applicable to safety cohort. | NA — The time frame is only applicable to safety cohort. | 0 | 1
  At day 190: Gastrointestinal disorders | NA — The time frame is only applicable to safety cohort. | NA — The time frame is only applicable to safety cohort. | NA — The time frame is only applicable to safety cohort. | 1 | 1
  At day 190: IPPC | NA — The time frame is only applicable to safety cohort. | NA — The time frame is only applicable to safety cohort. | NA — The time frame is only applicable to safety cohort. | 2 | 0
  At day 190: RTMD | NA — The time frame is only applicable to safety cohort. | NA — The time frame is only applicable to safety cohort. | NA — The time frame is only applicable to safety cohort. | 0 | 1
  At day 190: NBMU | NA — The time frame is only applicable to safety cohort. | NA — The time frame is only applicable to safety cohort. | NA — The time frame is only applicable to safety cohort. | 2 | 0
  At day 190: Social circumstances | NA — The time frame is only applicable to safety cohort. | NA — The time frame is only applicable to safety cohort. | NA — The time frame is only applicable to safety cohort. | 1 | 0

14. Primary Outcome: Number of Subjects With Signs of Long-Term Radiation Toxicity
Description: Long-term radiation toxicity included incidence of potential late toxicity, such as new primary cancers and bone marrow changes (acute myelogenous leukemia, myelodysplastic syndrome, and aplastic anemia).
Time Frame: From start of study treatment upto 12 months
Population: Only participants who received treatment were assessed
Measure: Number; unit: Participants
Arm/Group | Alpharadin 50 kBq/kg + Docetaxel 60 mg/m^2 - Safety Cohort | Docetaxel 75 mg/m^2 - Safety Cohort
Number analyzed (Participants) | 33 | 13
Participants | 2 | 0

15. Other Pre Specified Outcome: Exploratory Efficacy: Weighted Mean Area Under the Curve for Bone Turnover Biomarkers
Description: Weighted mean area under the curve for the below bone turnover biomarkers were evaluated, ICTP = pyridinoline cross-linked carboxyterminal telopeptide P1NP = N-terminal peptide of procollagen type 1 uCTX-1 = urine C-telopeptide 1
Time Frame: From start of study treatment to 6 weeks after study treatment (maximum 12 weeks in dose escalation; 30 weeks in the expanded safety cohort)
Population: Subjects included in the per protocol: All subjects in the ITT population who received at least 40% of the specified number of administrations of radium-223 dichloride (in the radium-223 dichloride cohort) or of docetaxel (in the docetaxel cohort), and who did not have any major protocol violations.
Measure: Mean (Standard Deviation); unit: mcg/L
Arm/Group | Alpharadin 50 kBq/kg + Docetaxel 60 mg/m^2 - Safety Cohort | Docetaxel 75 mg/m^2 - Safety Cohort
Number analyzed (Participants) | 32 | 13
mcg/L
  uCTX-1 | 14 (16.86) | 22.6 (28.2)
  P1NP | 42.9 (42.36) | 106.5 (118.93)
  ICTP | 4.7 (2.43) | 7 (7.08)

16. Other Pre Specified Outcome: Exploratory Efficacy: Time to Prostate-specific Antigen (PSA) Progression
Description: Serum PSA progression defined as two consecutive increases in PSA over a previous reference value within 6 months of first study treatment, each measurement at least 1 week apart.
Time Frame: 12 months
Population: as for outcome 15
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Alpharadin 50 kBq/kg + Docetaxel 60 mg/m^2 - Safety Cohort | Docetaxel 75 mg/m^2 - Safety Cohort
Number analyzed (Participants) | 32 | 13
days | 200 [175 to 278] | 146 [86 to 169]

17. Other Pre Specified Outcome: Exploratory Efficacy: Percent Change From Baseline in Circulating Tumor Cells at Day 85
Description: CTCs were measured to follow the evolution of the level of CTCs after treatment.
Time Frame: Baseline, Day 85, expanded safety cohort
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Alpharadin 50 kBq/kg + Docetaxel 60 mg/m^2 - Safety Cohort | Docetaxel 75 mg/m^2 - Safety Cohort
Number analyzed (Participants) | 32 | 13
Percent Change | -75.3 (55.29) | -68.4 (61.4)

18. Other Pre Specified Outcome: Exploratory Efficacy: Time to Clinical or Radiographic Progression
Description: Time to first radiologic or clinical progression is determined by one of the following:
  * For soft tissue lesions, the determination is based on Response Evaluation Criteria in Solid Tumors 1.1.
  * For bone disease, the determination is based on Prostate Cancer Working Cohort 2 (PCWG2) definitions, which require the appearance of at least 2 new lesions with a confirmatory bone scan at least 6 or more weeks later. For clinical progression, the investigators followed the recommendations of the PCWG25 and used their clinical judgment to determine clinical progression.
Time Frame: From start of study treatment to 12 months, at every 12 weeks
Population: as for outcome 15
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Alpharadin 50 kBq/kg + Docetaxel 60 mg/m^2 - Safety Cohort | Docetaxel 75 mg/m^2 - Safety Cohort
Number analyzed (Participants) | 32 | 13
days | 365 [248 to 372] | 284 [96 to 372]

19. Other Pre Specified Outcome: Progression Free Survival (PFS) End Point
Description: PFS defined as the time from randomization (randomization referred to the date of treatment assignment) to disease progression (radiological or clinical, whichever was earlier) or death (if death occurred before progression was documented). Subjects without progression or death at the time of analysis were censored at their last date of tumor evaluation.
Time Frame: From start of study treatment to 12 months, at every 12 weeks
Population: as for outcome 15
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Alpharadin 50 kBq/kg + Docetaxel 60 mg/m^2 - Safety Cohort | Docetaxel 75 mg/m^2 - Safety Cohort
Number analyzed (Participants) | 32 | 13
days | 189 [85 to 267] | 146 [86 to 169]

20. Other Pre Specified Outcome: Overall Survival Rate
Description: The overall survival (OS) time in days was calculated as number of days since the day of first dose of study medication until the date of death.
Time Frame: 12 months
Population: as for outcome 15
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Alpharadin 50 kBq/kg + Docetaxel 60 mg/m^2 - Safety Cohort | Docetaxel 75 mg/m^2 - Safety Cohort
Number analyzed (Participants) | 32 | 13
days | 89.1 [69.8 to 96.4] | 90 [47.3 to 98.5]

21. Other Pre Specified Outcome: Number of Subjects Who Responded to Interactive Voice Response System (IVRS) Pain
Description: The subject completed the full BPI (short form) paper questionnaire, and clinical staff completed the analgesic log. The test consists of 10 questions addressing severity, location, chronicity, and amount of relief. In question 3, subjects with pain are asked to evaluate the severity of pain at worst in the past 24 hours in a 0 to 10 scale, with 0 indicating no pain, and 10 indicating the worst pain.
Time Frame: From start of study treatment until 12 months
Population: as for outcome 15
Measure: Number; unit: Participants
Arm/Group | Alpharadin 50 kBq/kg + Docetaxel 60 mg/m^2 - Safety Cohort | Docetaxel 75 mg/m^2 - Safety Cohort
Number analyzed (Participants) | 32 | 13
Participants
  Day 1 | 23 | 11
  Day 22 | 24 | 11
  Day 43 | 22 | 10
  Day 64 | 21 | 10
  Day 85 | 20 | 11
  Day 106 | 20 | 9
  Day 127 | 19 | 6
  Day 148 | 18 | 5
  Day 169 | 17 | 5
  Day 190 | 17 | 5
  Safety Follow-up | 18 | 9
  6-Month Follow-up | 1 | 2
  9-Month Follow-up | 12 | 7
  12-Month Follow-up | 7 | 5

ADVERSE EVENTS:
Description: Number of participants at risk are from safety analysis set, please refer to participant flow section.
Groups:
- Alpharadin 25 kBq/kg + Docetaxel 75 mg/m^2 - Dose Escalation: Subjects received two intravenous injections of Alpharadin (Radium [Ra]-223 dichloride, BAY88-8223) at a dose of 25 kBq/kg body weight based on National Institute of Standards and Technology (NIST) 2010 standardization, separated by an interval of six weeks in combination with docetaxel at 75 milligram per square meter (mg/m^2) every three weeks; unless dose limiting toxicity (DLT) or other safety concerns limited the dose escalation
Arm/Group | Alpharadin 25 kBq/kg + Docetaxel 75 mg/m^2 - Dose Escalation | Alpharadin 25 kBq/kg + Docetaxel 60 mg/m^2 - Dose Escalation | Alpharadin 50 kBq/kg + Docetaxel 60 mg/m^2 - Dose Escalation | Alpharadin 50 kBq/kg + Docetaxel 60 mg/m^2 - Safety Cohort | Docetaxel 75 mg/m^2 - Safety Cohort
Serious Adverse Events (participants affected / at risk) | 4/7 | 0/3 | 2/7 | 7/33 | 4/13
Other Adverse Events (participants affected / at risk) | 7/7 | 3/3 | 7/7 | 33/33 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alpharadin 25 kBq/kg + Docetaxel 75 mg/m^2 - Dose Escalation (N=7) | Alpharadin 25 kBq/kg + Docetaxel 60 mg/m^2 - Dose Escalation (N=3) | Alpharadin 50 kBq/kg + Docetaxel 60 mg/m^2 - Dose Escalation (N=7) | Alpharadin 50 kBq/kg + Docetaxel 60 mg/m^2 - Safety Cohort (N=33) | Docetaxel 75 mg/m^2 - Safety Cohort (N=13)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (3) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blindness unilateral (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Biopsy lymph gland (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alpharadin 25 kBq/kg + Docetaxel 75 mg/m^2 - Dose Escalation (N=7) | Alpharadin 25 kBq/kg + Docetaxel 60 mg/m^2 - Dose Escalation (N=3) | Alpharadin 50 kBq/kg + Docetaxel 60 mg/m^2 - Dose Escalation (N=7) | Alpharadin 50 kBq/kg + Docetaxel 60 mg/m^2 - Safety Cohort (N=33) | Docetaxel 75 mg/m^2 - Safety Cohort (N=13)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (3) | 2 (2) | 5 (5) | 10 (28) | 5 (5)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 2 (3)
Ocular hypertension (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Anorectal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (3) | 11 (14) | 5 (6)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 2 (4) | 5 (5) | 14 (36) | 5 (9)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (4)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (4) | 1 (2) | 2 (3) | 16 (33) | 8 (13)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (7) | 2 (2)
Tongue ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0) | 2 (3) | 5 (9) | 2 (3)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 8 (24) | 2 (2)
Chest discomfort (General disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Facial pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 5 (5) | 3 (3) | 4 (4) | 17 (29) | 9 (15)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucosal dryness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 5 (5) | 2 (3)
Oedema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (7) | 1 (2)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 12 (16) | 5 (9)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Pyrexia (General disorders) | 1 (3) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatomegaly (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Herpes virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Oral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Rectal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tinea pedis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (2)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Radiation proctitis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2)
Respiratory rate increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 11 (13) | 4 (6)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Insulin resistance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 7 (9) | 6 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (2) | 1 (1) | 12 (16) | 4 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 2 (2)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (5)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 8 (9) | 2 (2)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 2 (2)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 7 (10) | 8 (12)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (5)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Myoclonus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 10 (12) | 4 (5)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 3 (4) | 0 (0) | 6 (8) | 2 (3)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Visual field defect (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 2 (2)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Nocturia (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 5 (6) | 0 (0)
Ureteric obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urethral pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Penile pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Priapism (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (5) | 3 (3)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 3 (3) | 2 (2) | 5 (5)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 3 (3) | 12 (12) | 7 (7)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (4)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nail bed disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 2 (2)
Nail dystrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 1 (2)
Nail toxicity (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 2 (2)
Skin atrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin striae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vascular pain (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The radium 223 dichloride treatment was calculated as 50 kBq per NIST 2010, and would be approximately 55 kBq per NIST 2015 standard. Pharmacokinetic endpoint was deleted as no PK variables were evaluated in the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less